CLINICAL TRIAL: NCT01741597
Title: A First Time in Human Phase I Imaging Study of iRGD in Patients With Advanced Breast and Pancreas Cancer
Brief Title: Dynamic Contrast Enhanced MRI in Patients With Advanced Breast or Pancreatic Cancer With Metastases to the Liver or Lung
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI chose to close the study
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12228; NCI-2012-02449 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA043904 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Liver Metastases; Lung Metastases; Recurrent Breast Cancer; Recurrent Pancreatic Cancer; Stage IV Breast Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms | interventions — N-end cysteine peptide tumor-homing peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (DCE-MRI, tumor-homing peptide iRGD) (Experimental): Patients undergo DCE-MRI on day 1 and undergo tumor-homing peptide iRGD DCE-MRI on day 2.
  Interventions: Procedure: dynamic contrast-enhanced magnetic resonance imaging; Other: pharmacological study; Biological: tumor-homing peptide iRGD

INTERVENTIONS:
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Undergo DCE-MRI
  Other Names: DCE-MRI
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Biological: tumor-homing peptide iRGD — Undergo tumor-homing peptide iRGD DCE-MRI
  Other Names: iRGD

SUMMARY:
This phase I trial studies the side effects of dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) in patients with advanced breast or pancreatic cancer with metastases to the liver or lung. Diagnostic procedures, such as DCE-MRI, may help measure a patient's response to treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the ability of iRGD (tumor-homing peptide iRGD) to elicit changes in metastatic breast cancer vascular permeability as measured by dynamic contrast enhanced (DCE) MRI.

II. To evaluate the pharmacokinetics of iRGD. III. To explore the safety of iRGD.

SECONDARY OBJECTIVES:

I. To explore changes in water diffusion status in tumors due to iRGD as measured by diffusion-weighted (DWI) MRI.

II. To explore the ability of iRGD to elicit changes in primary pancreatic cancer vascular permeability as measured by dynamic contrast enhanced (DCE) MRI.

III. To explore changes in water diffusion status in primary pancreatic cancer due to iRGD as measured by DWI-MRI.

OUTLINE:

Patients undergo DCE-MRI on day 1 and undergo tumor-homing peptide iRGD DCE-MRI on day 2.

After completion of study treatment, patients are followed up for 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologic diagnosis of breast or pancreatic adenocarcinoma (expansion cohort) metastatic to the liver or lung
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Women of child-bearing potential must have a negative serum pregnancy test within 7 days of the first DCE-MRI and must have agreed to use an effective contraceptive method; the effects of iRGD on the developing fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Patient must have a measurable lesion at least 2 cm in size amenable to DCE-MRI study as determined by Radiology
* Computed tomography (CT)/MRI scan must be obtained within 3 weeks prior to study entry
* Absolute neutrophil count >= 1,500/mcl
* Platelet count >= 100,000/mcl
* Creatinine =< 1.3 mg/dl or a measured creatinine clearance >= 60 cc/min
* Bilirubin =< 1.5 mg/dl
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) no greater than 2.5 times the upper limit of normal for patients with liver metastases; patients without liver metastasis should have ALT and AST no greater than 1.5 times the upper limit of normal
* Patients currently being treated for severe infections or who are recovering from major surgery or other intercurrent illnesses are ineligible until recovery is deemed complete by the investigator
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Patients with grade 2 or higher toxicity due to previous chemotherapy; all toxicities should recover to grade 0 or 1 prior to day 1

Exclusion Criteria:

* Patients experiencing an infusion reaction with the day 1 DCE-MRI
* Patients with any grade electrolyte abnormalities that are unable to be corrected by day 1
* Patients with a history of previous reaction to IV contrast
* Impaired cardiac function including any one of the following:

  * Complete left bundle branch block or use of a permanent cardiac pacemaker
  * Congenital long QT syndrome
  * Presence of ventricular tachyarrhythmias
  * Clinically significant resting bradycardia (< 50 beats per minute)
  * Corrected Fridericia's QT interval (QTcF) > 450 msec on screening electrocardiogram (ECG)
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
* Presence of atrial fibrillation
* Previous history angina pectoris or acute myocardial infarction (MI) within 6 months
* Congestive heart failure (New York Heart Association functional classification III-IV)
* Uncontrolled hypertension (mmHg > 140 systolic or > 90 diastolic)
* Brain or leptomeningeal metastases
* Patients with an active, bleeding diathesis or requiring therapeutic anticoagulation
* Patients receiving bevacizumab within 3 months of study entry
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients should not have any uncontrolled illness including ongoing or active infection
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to iRGD
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in volume transfer coefficient (Ktrans) during DCE-MRI with tumor-homing peptide iRGD compared to a baseline DCE-MRI without tumor-homing peptide iRGD | Baseline to 15 days
  Analyzed using a multi-compartment pharmacokinetic modeling algorithm already implemented at multiple clinical trial sites for breast and body imaging.

SECONDARY OUTCOMES:
The potential for tumor-homing peptide iRGD to enhance uptake of key anti-cancer agents | Up to 15 days
  Analyzed using a multi-compartment pharmacokinetic modeling algorithm already implemented at multiple clinical trial sites for breast and body imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States